CLINICAL TRIAL: NCT05050786
Title: Prophylactic Negative-Pressure Wound Treatment (NPWT) for Patients Undergoing Elective Open Incisional Hernia Repair: the PROPRESS Trial
Brief Title: Prophylactic Negative Pressure Wound Therapy for Patients Undergoing Incisional Hernia Repair
Acronym: PROPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kristian Kiim Jensen (Other)
Responsible Party: Sponsor-Investigator, Kristian Kiim Jensen, MD, PHD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PROPRESS
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Incisional Hernia; Surgical Wound Infection; Surgical Site Infection; Quality of Life
Keywords: negative wound pressure therapy; incisional hernia repair; closed incision; randomized clinical trial; surgical site infection; surgical wound infection
MeSH Terms: conditions — Incisional Hernia; Surgical Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard wound dressing (Active Comparator)
  Interventions: Other: Standard Wound Dressing
- Negative Pressure Wound Therapy (NPWT) (Experimental)
  Interventions: Device: Negative Wound Pressure Therapy (Prevena(TM))

INTERVENTIONS:
Device: Negative Wound Pressure Therapy (Prevena(TM)) — After skin closure, NPWT in the form of Prevena™ (KCI/Acelity, San Antonia, TX, USA) is applied using the following technique: The sterile foam dressing is removed from the package and placed on the incision in the entire length, on top of which the sterile dressing is placed, ensuring air tightness. An appropriate hole in the dressing is cut at the center of the dressing and the tube for the interface pad is connected and a negative pressure of 125mmHg is applied. The Prevena™ system is removed on the morning of postoperative day 3.
  Arms: Negative Pressure Wound Therapy (NPWT)
Other: Standard Wound Dressing — After skin closure, a standard operative dressing is applied in the entire length of the incision. This operative dressing is removed in the morning of postoperative day two. Only in the case of blood or serous fluid mandating changing of the dressing, will this be done prior to postoperative day 2.
  Arms: Standard wound dressing

SUMMARY:
The study will examine the effect of using Negative Pressure Wound Therapy (NPWT) compared with standard wound dressing among patients undergoing elective open surgery for incisional hernia. The study's main hypothesis is that NPWT will decrease the post-operative incidence of surgical site infections and also improve the patients' quality of life including less scar-related pain and higher cosmetic satisfaction.

DETAILED DESCRIPTION:
In recent years, negative pressure wound therapy (NPWT) has been utilized for the treatment of complicated wounds within orthopedic and vascular surgery, whereas incisions after abdominal surgery have not been treated with prophylactic negative pressure wound treatment to the same extent. Patients undergoing incisional hernia repair per definition have elicited insufficient wound healing (i.e. the hernia), and often carry comorbidities such as diabetes, obesity and a history of smoking, leaving them at a high risk of developing wound complications. Despite efforts to reduce this risk, the incidence remains as high as 50% in some series. Wound complications are especially concerning in patients undergoing incisional hernia repair, as a foreign body (synthetic polypropylene mesh) is placed in the abdominal wall during the procedure. Wound complications are directly associated with an increased risk of hernia recurrence, which reduces the patients' quality of life and has severe socioeconomic costs including a higher risk of prolonged hospital admission, re-operation, re-admission and increased mortality (2). The aim of this trial is to examine the effects of prophylactic NPWT on postoperative wound complications after open incisional hernia repair compared with standard care, i.e. an operative dressing. It is our hypothesis that NPWT significantly reduces the incidence of surgical site infections (SSI) as defined by the Center for Disease Control.

Since Bispebjerg Hospital in Denmark is the regional center for complex hernias, this is one of the few sites where a randomized trial including 110 patients undergoing open incisional hernia repair is feasible. To date, only five randomized controlled trials of prophylactic NPWT for closed abdominal incisions have been published. In the most recent meta-analysis of these trials, there was no reduced risk of wound complications in patients treated with NPWT, however results indeed seemed subjective to type-II error (relative risk 0.56 (95% confidence interval 0.30-1.03, P = 0.064). Thus, adding another randomized trial expectedly will alter the conclusion of the next meta-analysis.

The study type is a randomized controlled trial (RCT) comprising two treatment groups, i.e. one of the following:

1. STANDARD CARE After skin closure, a standard operative dressing is applied in the entire length of the incision. This operative dressing is removed in the morning of postoperative day two. Only in the case of blood or serous fluid mandating changing of the dressing, will this be done prior to postoperative day 2.
2. INTERVENTION After skin closure, NPWT in the form of Prevena™ (KCI/Acelity, San Antonia, TX, USA) is applied using the following technique: The sterile foam dressing is removed from the package and placed on the incision in the entire length, on top of which the sterile dressing is placed, ensuring air tightness. An appropriate hole in the dressing is cut at the center of the dressing and the tube for the interface pad is connected and a negative pressure of 125mmHg is applied. The Prevena™ system is removed on the morning of postoperative day 3.

Patients are included in the study during the planning of surgery in the outpatient clinic or within a week before surgery at the planned visit in the department of surgery. Patients are randomized to intervention or standard treatment in a 1:1 allocation ratio, which will be performed using computer generated sequences with varying block sizes (http://www.sealedenvelope.com/). This randomization will generate randomization and code envelopes and is carried out by a physician not otherwise involved in the study. On the day of surgery, the patients are given a randomization number. Corresponding randomization envelopes contain information about the intervention the patient is to receive and are thus opened during surgery, i.e. immediately after closure of the linea alba, whereas the code envelopes will be opened at the time of data analysis after all included patients have completed 30-day follow up. Based on the average number of elective open incisional hernia repairs at the study's operating site, the patient recruitment is expected to take 1 to 2 years.

PARTICIPANTS

The following baseline data are registered for each participant:

* Age [nominal: number]
* Sex [categorical: Male, Female]
* Number of previous abdominal operations [nominal: number]
* Number of previous incisional hernia repairs [nominal: number]
* Smoking status [categorical: Active smoker, Non-smoker]
* BMI [kg/m2]
* Chronic obstructive pulmonary disease [categorical: Yes, No]
* Diabetes [categorical: Yes, No]
* American Society of Anesthesiology (ASA) class [categorical: 1, 2, 3, 4, 5]
* Site of incisional hernia [categorical: Midline, Upper left, Lower left, Upper right, Lower right, Other]
* Orientation of hernia incision [categorical: Horizontal, Vertical]
* Bleeding disorder + anticoagulative medication [categorical: Yes, No]
* Serum albumin level [numerical: g/L]
* Maximal horizontal fascial defect [numerical: centimeters]
* Maximal vertical fascial defect [numerical: centimeters]
* Botox [categorical: Yes, No]

Perioperative established variables

* Type of procedure/repair [categorical: Rives-Stoppa, RS+TAR, onlay, IPOM, RS+ECS, other]
* Operative time [numerical: minutes]
* Length of incision [numerical: centimeters]
* Contamination grade [categorical: clean, clean-contaminated, contaminated, dirty]
* Type of mesh
* Commentary option (e.g. perioperative complications)

ETHICAL CONSIDERATIONS This trial aim to improve the treatment of patients undergoing open abdominal surgery by reducing the incidence of wound complications. We hypothesize that the intervention will be an improvement compared with the standard treatment currently offered, without any severe side-effects. This includes both in terms of the expected reduction in wound complication incidence as well as an increase in patient quality of life. Thus, the expected benefits from participation in the current trials outweigh any potential drawbacks and is therefore considered ethical appropriate. Lastly, the trial conforms to the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective open incisional hernia repair

Exclusion Criteria:

* active superficial or deep wound infection
* inability to provide informed consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | The outcome will be monitored over a 30 days period post surgery. The patient is typically discharged on day 3 and will be notified of signs of infection by standard including warning signs that should lead to medical contact.
  As defined by the Center for Disease Control

SECONDARY OUTCOMES:
Pooled Incidence of Surgical Site Occurence | This will be evaluated at the 30 day follow up contact
  Surgical site infection, wound hematoma, skin necrosis or superficial wound dehiscence
Patient-reported pain and satisfaction with the scar at 30-day follow-up | This will be evaluated at the 30 day follow up contact
  Standardized questionnaire POSAS
Patient-reported Hernia-related Quality of life score at 30-day follow-up | This will be evaluated at the 30 day follow up contact
  Standardized questionnaire EuraHS-QoL

CONTACTS AND LOCATIONS:
Overall Officials: Mads Marckmann, MD, Principal Investigator — Digestive Disease Center, Bispebjerg Hospital, Denmark
Locations (1):
- Kristian Schaumburg Kiim, Copenhagen NV, Copenhagen, Denmark

REFERENCES:
- [Background] Kaoutzanis C, Leichtle SW, Mouawad NJ, Welch KB, Lampman RM, Wahl WL, Cleary RK. Risk factors for postoperative wound infections and prolonged hospitalization after ventral/incisional hernia repair. Hernia. 2015 Feb;19(1):113-23. doi: 10.1007/s10029-013-1155-y. Epub 2013 Sep 13. PMID 24030572
- [Background] Badia JM, Casey AL, Petrosillo N, Hudson PM, Mitchell SA, Crosby C. Impact of surgical site infection on healthcare costs and patient outcomes: a systematic review in six European countries. J Hosp Infect. 2017 May;96(1):1-15. doi: 10.1016/j.jhin.2017.03.004. Epub 2017 Mar 8. PMID 28410761
- [Background] Li PY, Yang D, Liu D, Sun SJ, Zhang LY. Reducing Surgical Site Infection with Negative-Pressure Wound Therapy After Open Abdominal Surgery: A Prospective Randomized Controlled Study. Scand J Surg. 2017 Sep;106(3):189-195. doi: 10.1177/1457496916668681. Epub 2016 Sep 8. PMID 27609528
- [Background] Shen P, Blackham AU, Lewis S, Clark CJ, Howerton R, Mogal HD, Dodson RM, Russell GB, Levine EA. Phase II Randomized Trial of Negative-Pressure Wound Therapy to Decrease Surgical Site Infection in Patients Undergoing Laparotomy for Gastrointestinal, Pancreatic, and Peritoneal Surface Malignancies. J Am Coll Surg. 2017 Apr;224(4):726-737. doi: 10.1016/j.jamcollsurg.2016.12.028. Epub 2017 Jan 11. PMID 28088597
- [Background] Kuper TM, Murphy PB, Kaur B, Ott MC. Prophylactic Negative Pressure Wound Therapy for Closed Laparotomy Incisions: A Meta-analysis of Randomized Controlled Trials. Ann Surg. 2020 Jan;271(1):67-74. doi: 10.1097/SLA.0000000000003435. PMID 31860549
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Soares KC, Baltodano PA, Hicks CW, Cooney CM, Olorundare IO, Cornell P, Burce K, Eckhauser FE. Novel wound management system reduction of surgical site morbidity after ventral hernia repairs: a critical analysis. Am J Surg. 2015 Feb;209(2):324-32. doi: 10.1016/j.amjsurg.2014.06.022. Epub 2014 Aug 7. PMID 25194761
- [Background] Kobayashi M, Mohri Y, Inoue Y, Okita Y, Miki C, Kusunoki M. Continuous follow-up of surgical site infections for 30 days after colorectal surgery. World J Surg. 2008 Jun;32(6):1142-6. doi: 10.1007/s00268-008-9536-6. PMID 18338205
- [Background] Javed AA, Teinor J, Wright M, Ding D, Burkhart RA, Hundt J, Cameron JL, Makary MA, He J, Eckhauser FE, Wolfgang CL, Weiss MJ. Negative Pressure Wound Therapy for Surgical-site Infections: A Randomized Trial. Ann Surg. 2019 Jun;269(6):1034-1040. doi: 10.1097/SLA.0000000000003056. PMID 31082899
- [Background] O'Leary DP, Peirce C, Anglim B, Burton M, Concannon E, Carter M, Hickey K, Coffey JC. Prophylactic Negative Pressure Dressing Use in Closed Laparotomy Wounds Following Abdominal Operations: A Randomized, Controlled, Open-label Trial: The P.I.C.O. Trial. Ann Surg. 2017 Jun;265(6):1082-1086. doi: 10.1097/SLA.0000000000002098. PMID 27926575
- [Derived] Marckmann M, Henriksen NA, Krarup PM, Helgstrand F, Vester-Glowinski P, Christoffersen MW, Kiim KS. Effect of standard wound dressing versus prophylactic closed incision negative-pressure therapy on surgical-site infection after open incisional hernia repair: multicentre randomized clinical trial. Br J Surg. 2025 Nov 29;112(12):znaf230. doi: 10.1093/bjs/znaf230. PMID 41316999
- See also: Definition of Surgical Site Infection (SSI) on page 10 — https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
- See also: Website for generating sequences with varying block sizes for randomization — http://www.sealedenvelope.com/